CLINICAL TRIAL: NCT04675775
Title: Medically-Tailored Meals to Prevent Recurrent Hepatic Encephalopathy: The BRAINFOOD Pilot Trial
Brief Title: The BRAINFOOD Trial to Prevent Recurrent Hepatic Encephalopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elliot B. Tapper, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00168821; P30AG024824 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Cirrhosis; Ascites; Liver Diseases; Frailty; Sarcopenia; Hepatic Encephalopathy
Keywords: Nutrition
MeSH Terms: conditions — Fibrosis; Ascites; Liver Diseases; Frailty; Sarcopenia; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medically-tailored meals (Experimental): Participants will receive meals that adhere to their specified nutritional targets dependent upon their cirrhosis complication of hepatic encephalopathy (HE) and/or ascites. Participants with HE will receive high-protein (approximately 1 gram of medication per kilogram of the body weight (1g/kg/day) and high-calorie (approximately 30c/kg/day) meals. Participants with HE and ascites will receive high-protein and high-calorie meals that are also low-sodium (less than or equal to 2000 milligrams a day).
  Interventions: Other: Medically-tailored meals (MTM); Dietary Supplement: Protein supplements; Behavioral: Nutrition education handout

INTERVENTIONS:
Other: Medically-tailored meals (MTM) — After the run-in baseline period participants will be expected to consume the meals and protein supplements meals between approximately Weeks 4 - 11 of the study. Additionally, participants will complete surveys before, during and after the meals.
Dietary Supplement: Protein supplements — A daytime and nighttime protein supplement will be provided after the baseline visit and should be consumed daily at home during the same study days as MTM. The daytime protein supplement is a protein bar (ZonePerfect or Perfect Bar). The nighttime supplement is a protein powder or liquid that can be dissolved in either water or milk.
  This is provided to participants with ProCel Vanilla Whey Protein powder which provides 15 grams of protein per serving or the ProCel LiquaCel liquid protein supplement mango, grape, watermelon and/or lemon flavors which provides 16g of protein per serving.
Behavioral: Nutrition education handout — A standardized nutrition education handout containing instructions on following a high-protein and sodium restricted diet (depending on the presence of ascites) will be given as part of Standard of Care.

SUMMARY:
This study is being completed for patients with cirrhosis, including patients with a prior history of hepatic encephalopathy (HE) to evaluate the feasibility and benefits of medically-tailored meals as an intervention.

Patients will be enrolled from the University of Michigan and will complete the baseline assessments in-person or remotely. In addition participants will complete study related materials before, during and after treatment with medically-tailored meals (MTM). After completing the study meals, participants will return for follow-up or have this visit completed remotely as well as have an observational period for 12 more weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis will be based upon:

  1. liver biopsy, OR
  2. history of cirrhosis complication: ascites, variceal bleeding, hepatic encephalopathy, OR
  3. 2 of the following 4 criteria:

     1. Ultrasound, Computed tomography (CT), or Magnetic resonance imaging (MRI) findings of cirrhosis (cirrhotic appearing liver, splenomegaly, varices, ascites)
     2. Fibroscan liver stiffness score >13 kilopascals (kPa)
     3. Laboratory testing: aspartate aminotransferase/platelet ratio index (APRI) >2.0
     4. CT, MRI or esophagogastroduodenoscopy (EGD) showing presence of esophageal varices
* Patients with history of > grade 2 HE within 180 days of enrollment based on review of clinical documentation verifying the event. If a description of HE symptoms is provided in clinical documentation, but it is unclear if it meets Grade 2 criteria, the principal investigator will assess the clinical documentation and provide an HE grade.

Exclusion Criteria:

* Non-English speaking
* Model for End-Stage Liver Disease (MELD) Score > 20
* Pregnancy (self-reported)
* Unable or unwilling to provide consent
* History of liver transplant
* Current or planned admission to a nursing facility
* Serum creatinine > 2.0 milligrams per deciliter (mg/dL) (with the exception that we will include patients with a serum creatinine > 2.0 mg/dL if they are receiving hemodialysis)
* Disorientation at the time of enrollment
* Barcelona-Clinic Liver Cancer (BCLC) Stage D Hepatocellular Carcinoma with Child-Turcotte-Pugh (CTP) Class C
* History of eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Medically-tailored Meals: Participants will receive meals that adhere to their specified nutritional targets dependent upon their cirrhosis complication of hepatic encephalopathy (HE) and/or ascites. Participants with HE will receive high-protein (approximately 1 gram of medication per kilogram of the body weight (1g/kg/day) and high-calorie (approximately 30c/kg/day) meals. Participants with HE and ascites will receive high-protein and high-calorie meals that are also low-sodium (less than or equal to 2000 milligrams a day).
  Medically-tailored meals (MTM): After the run-in baseline period participants will be expected to consume the meals and protein supplements meals between approximately Weeks 4 - 11 of the study. Additionally, participants will complete surveys before, during and after the meals.
  Protein supplements: A daytime and nighttime protein supplement will be provided after the baseline visit and should be consumed daily at home during the same study days as MTM. The daytime protein supplement is a protein bar (ZonePerfect or Perfect Bar). The nighttime supplement is a protein powder or liquid that can be dissolved in either water or milk.
  This is provided to participants with ProCel Vanilla Whey Protein powder which provides 15 grams of protein per serving or the ProCel LiquaCel liquid protein supplement mango, grape, watermelon and/or lemon flavors which provides 16g of protein per serving.
Period: Overall Study
Arm/Group | Medically-tailored Meals
Started | 17
Participants Who Did Not Withdraw Prior to MTM | 12
Participants Who Did Not Withdraw During MTM | 10
Completed | 10
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: 17 participants total were enrolled. Of those 17, 5 withdrew from the trial before receiving the medically-tailored meals (MTM), and 2 more withdrew during the trial. The data from the 7 participants who withdrew was not used in the results. The baseline data presented below is only for the participants who completed the trial.
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 59.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Non-white | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Retention Rate Based on Proportion of Participants Who Complete All Study Visits
Description: Overall participant retention rate based on proportion of participants who completed all study visits
Time Frame: up to 27 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 17
Participants | 10

2. Primary Outcome: Participant Adherence Rate to Medically-Tailored Meals (MTM)
Description: The participant adherence rate to MTM based on proportion of participants who consumed ≥75% of delivered meals and evening snack
Time Frame: up to 11 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 17
Participants | 10

3. Secondary Outcome: Proportion of Participants Who Completed All Study Assessments and Procedures
Description: The number of participants who completed all study assessments and procedures during each study visit compared to the number of participants who did not complete all study assessments and procedures.
Time Frame: up to 27 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 10
Participants | 8

4. Secondary Outcome: Eligible Candidates Who Enrolled After Screening
Description: Results show the participants who enrolled in the trial following determination of the total number of candidates who were screened and determined to be eligible to participate in the trial.
Time Frame: approximately 1 year (enrollment period)
Population: 30 individuals who were screened were determined to meet the eligibility criteria for this trial. Of those 30, 10 declined to participate and 3 did not participate for other reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 30
Participants | 17

5. Secondary Outcome: The Percentage of Enrolled Participants Who Dropped Out of Study
Description: The percentage of enrolled participants who dropped out of either study stage before the final study visit due to withdrawal by participant or lost to follow-up, and not due to death, withdrawal by study staff or principal investigator discretion.
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 17
Participants | 7

6. Secondary Outcome: Time Required to Complete Assessments
Description: Feasibility of the assessments were evaluated by measuring the amount of time participants required to complete all assessments in minutes.
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Medically-tailored Meals
Number analyzed (Participants) | 17
minutes | 43.27 (21.44)

7. Other Pre Specified Outcome: The Proportion of Participants Who Complete All 24-hour Diet Recall Interviews
Description: The proportion of participants who complete all 24-hour Diet Recall interviews compared to the number of participants who did not complete all 24-Hour Diet Recall interviews.
Time Frame: up to 11 weeks post enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change is EncephalApp - Stroop Score
Description: This was a computerized, timed test of attention conducted on an Interactive Personal Application Device (iPad) or smart device by a phone application that asked participants to identify the color of words. The score was the sum of the time it took to complete color-word concordance and color-word discordance. A score of less than 190 was considered 'normal' cognitive function. Participants who were color-blind were excluded from performing this test.
Time Frame: baseline, up to 13 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in One Minute Animal Naming Test (ANT)
Description: The participants listed as many unique animals as possible in 60 seconds.
Time Frame: baseline, up to 27 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 27 weeks
Arm/Group | Medically-tailored Meals
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medically-tailored Meals (N=17)
Exacerbation of cirrhosis (Hepatobiliary disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04675775/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT04675775/ICF_001.pdf